CLINICAL TRIAL: NCT00803868
Title: Pilot Study of Varenicline (Chantix®) in the Treatment of Friedreich's Ataxia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The DSMB recommended that the study be stopped as a result of concerns regarding safety and intolerability and insufficient evidence of efficacy.
Sponsor: University of South Florida (Other)
Collaborators: Friedreich's Ataxia Research Alliance (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6
Record Dates: First submitted 2008-12-04; First posted 2008-12-08 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Varenicline
  Interventions: Drug: varenicline
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — up to 1mg po bid for 9 weeks
  Arms: 1
Drug: placebo — placebo matching study drug up to 1mg po bid
  Arms: 2

SUMMARY:
The purpose of this study is to determine if varenicline is effective in treating symptoms of Friedreich's ataxia.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with FA diagnosed by confirmed by genetic testing.
2. Age 18 years to 80 years.
3. Women who are not pregnant or breast feeding, and who do not intend to become pregnant. Women of child-bearing potential must use a reliable method of contraception and must provide a negative urine pregnancy test at entry into the study.
4. CBC, CMP, and diabetes lab results not indicative of clinically relevant abnormalities (results within the past 6 months prior to screening). These would include but are not limited to:

   Electrolytes (Chloride, Sodium, Potassium) within laboratory defined normal limits.

   Hemoglobin, white cell count, platelet count and fasting glucose within laboratory defined normal limits. Creatinine must be (≤1.5 mg/dl).

   ALT (6-40 u/l) and AST (10-30 u/l) must be less than 2 times normal limit
5. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
6. Patient permission (informed consent).
7. Ambulatory status: Half of the enrolled patients must be able to ambulate with or without assistance; half of the enrolled patients must be non-ambulatory.

Exclusion Criteria:

1. Any unstable illness that in the investigator's opinion preclude participation in this study.
2. Use of another investigational product within the past 28 days.
3. Patients with a history of substance abuse.
4. Presence of preexisting psychiatric illness (specifically schizophrenia, bipolar disorder, or history of suicide attempt).
5. Presence of diabetes (as determined by fasting blood glucose labs within the past 6 months).
6. Presence of clinically significant cardiac disease (as determined by the investigator based on EKG and echocardiogram results within the past 6 months). Specifically, patients with an ejection fraction <40% or a prolonged QT interval (>50% of cycle duration) will be excluded. If abnormalities are noted on the EKG or echocardiogram, the patient will be eligible IF they provide clearance from a cardiologist.
7. Presence of current uncontrolled depression as measured by PHQ9 (criteria for depression include all of the following to be present: At least one of the first two questions on PHQ9 endorsed as positive (little pleasure, feeling depressed) indicating the symptom has been present more than half the time in the past two weeks; Question 10 about difficulty at work or home or getting along with others should be answered at least "somewhat difficult."; and the total score ≥ 10.
8. Concurrent treatment with any MAOIs, Wellbutrin, or nicotine patches.
9. Patients who currently smoke or have smoked within the past 12 months (Smoking will be defined as having smoked any substance even on a single occasion).
10. Dementia or other psychiatric illness that prevents the patient from giving informed consent (MMSE less than 25).
11. Legal incapacity or limited legal capacity.
12. Presence of severe renal disease (creatinine >1.6) or hepatic disease (AST or ALT>2x times normal) (as evidenced by labs reported within the past 6 months).
13. Abnormal WBC hemoglobin or platelet count (as evidenced by labs reported within the past 6 months).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Friedreich Ataxia Rating Scale (FARS) | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, M.D., Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania